CLINICAL TRIAL: NCT00539903
Title: Physical Activity and Immigrant Health
Acronym: FAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 07112001326
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Physical Activity
Keywords: Activity Level
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator

INTERVENTIONS:
Behavioral: Physical activity (PA) and immigrants

SUMMARY:
There is today a growing need for culturally adapted initiatives among immigrants to prevent and treat T2D. Others have failed to increase the level of physical activity in this sedate group. The investigators believe this is due to missing assistance and lack of influence from the Pakistani milieu. To improve this, a culturally adapted physical activity will be established in this project in close cooperation with the Pakistanis themselves.

Through this program it is the investigators' goal to increase their physical activity level and prevent lifestyle diseases among Pakistanis in Oslo with a high risk of developing these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Pakistani background
* 25-55 year old
* Physically inactive

Exclusion Criteria:

* Diabetes
* heart condition
* medication that could affect the results

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2008-08

PRIMARY OUTCOMES:
Physical activity level

CONTACTS AND LOCATIONS:
Overall Officials: Eivind Andersen, MsC, Principal Investigator — Norwegian School of Sport Sciences
Locations (1):
- Norwegian school of sport sciences, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Andersen E, Burton NW, Anderssen SA. Physical activity levels six months after a randomised controlled physical activity intervention for Pakistani immigrant men living in Norway. Int J Behav Nutr Phys Act. 2012 Apr 26;9:47. doi: 10.1186/1479-5868-9-47. PMID 22537281